CLINICAL TRIAL: NCT05850585
Title: A Prospective, Double-blind, Randomized Controlled Trial of FMT Combined With Antipsychotic Drugs to Improve the Efficacy of Schizophrenia
Brief Title: A Study of the Efficacy of Fecal Microbiota Transplantation(FMT) in the Treatment of Schizophrenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 82022023-2; 2021GXLH-Z-083-2 (Other Grant/Funding Number: Key Research and Development Plan of Shaanxi Province)
Record Dates: First submitted 2023-04-12; First posted 2023-05-09 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbiota transplantation(FMT) (Experimental): Subjects will receive FMT capsules (10^12 Colony-Forming Units(CFU)/capsule) in addition to their usual antipsychotics treatment. Subjects will continue to receive FMT capsules for 8 weeks. During this period, both groups could receive first-line atypical antipsychotics recommended by current treatment guidelines.
  Interventions: Drug: Fecal microbiota transplantation(FMT)
- Placebo (Placebo Comparator): Participants will receive a placebo capsule with the same color, appearance, and smell as the FMT capsule, in addition to their usual antipsychotics treatment. Placebo capsules contained the food probiotic Lactobacillus (10^12 CFU per capsule). Subjects will continue to receive placebo capsules for 8 weeks. During this period, both groups could receive first-line atypical antipsychotics recommended by current treatment guidelines.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fecal microbiota transplantation(FMT) — Subjects will receive FMT capsules (10^12 Colony-Forming Units(CFU)/capsule) in addition to their usual antipsychotics treatment. Subjects will continue to receive FMT capsules for 8 weeks. During this period, both groups could receive first-line atypical antipsychotics recommended by current treatment guidelines.
  Arms: Fecal microbiota transplantation(FMT)
Other: Placebo — Participants will receive a placebo capsule with the same color, appearance, and smell as the FMT capsule, in addition to their usual antipsychotics treatment. Placebo capsules contained the food probiotic Lactobacillus (10^12 CFU per capsule). Subjects will continue to receive placebo capsules for 8 weeks. During this period, both groups could receive first-line atypical antipsychotics recommended by current treatment guidelines.
  Arms: Placebo

SUMMARY:
The purpose of this study was to explore whether repeated oral fecal capsules could improve outcomes in patients with schizophrenia receiving conventional antipsychotic drugs. This study was divided into screening period (1 week) and treatment period (8 weeks). Subjects who met the inclusion criteria during the screening period entered the treatment period. During the treatment period, the patients were divided into two groups: oral fecal bacteria capsules + antipsychotics group; Oral placebo + antipsychotic group. During the follow-up period, both groups were treated with stable dose of antipsychotic drugs during the treatment period. Before and after the intervention, venous blood samples of patients were collected for routine tests such as liver and kidney function to determine the safety of treatment. The scale evaluated the improvement of patients' psychotic symptoms to determine the efficacy and safety of FMT combined with antipsychotics.

DETAILED DESCRIPTION:
The main research content of this project is to observe the efficacy and safety of adjuvant FMT capsules in the treatment of schizophrenia by enrolling patients with schizophrenia and randomly administering FMT combined with antipsychotics or placebo combined with antipsychotics.

This is a multicenter, randomized, double-blind, placebo-controlled clinical trial. In this study, patients with schizophrenia were randomly divided into two groups. The first group was the experimental group, and FMT capsules (10^12 CFU/ capsule) were used in addition to conventional antipsychotic drugs. The other group, a control group, received a placebo pill with the same color, appearance and smell as the FMT capsules in addition to regular antipsychotic medication. Placebo capsules contain Lactobacillus probiotics for food use (10^12 CFU/ capsule). To observe the efficacy and safety of adjuvant FMT capsule in patients with schizophrenia.

The subjects (inpatients) were evaluated for meeting the eligibility requirements for this study according to the pre-specified inclusion and exclusion criteria, and demographic data (age, sex, marital status, educational level, employment, height and weight, smoking and drinking, and other general information as well as questionnaire assessment of eating habits) were collected. Improve laboratory examination (blood routine, liver function, kidney function and lipid), electrocardiogram and scale assessment.

Patients at the end of the screening period were randomly assigned to the experimental and control groups. Subjects will continue to receive FMT capsules or placebo capsules until the end of 8 weeks. During this period, both groups were given first-line atypical antipsychotics (clozapine, olanzapine, quintiapine, risperidone, aripiprazole, Ziprasidone, amsulapride, paliperidone, and paliperidone palmitate) recommended by current treatment guidelines, and added to the effective therapeutic dose within 1 week.

Benzodiazepines and drugs that ameliorate side effects of antipsychotics may be used during the study period. Antidepressants and mood stabilizers are prohibited. Transcranial magnetic stimulation and electronic biofeedback were allowed during the study, and non-convulsive electroconvulsive therapy was prohibited.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 65 years
* Patients with schizophrenia and a disease duration of 5 years or less are currently receiving first-line recommended antipsychotic medications
* The patients met the diagnostic criteria of schizophrenia in the 10th edition of the International Classification of Diseases (ICD-10)
* Positive and Negative Syndrome Scale (PANSS) : total score ≥60 (at least 3 positive items ≥3 or 3 negative items ≥3)
* Junior high school or above
* Subjects provided informed consent

Exclusion Criteria:

* Pregnant and lactating women
* Clinically significant or unstable medical diseases, including congestive heart failure, liver and kidney failure, cancer, immune and metabolic endocrine diseases
* Or hepatobiliary gastrointestinal diseases, abdominal pain, diarrhea (except functional constipation)
* Those who had acute or chronic infection, had taken anti-inflammatory drugs, cortisol hormones, and had received antibiotics in the past month
* Other neuropsychiatric disorders (patients with organic brain lesions, mental disorders and mental retardation caused by physical diseases or psychoactive substances)
* There were those with fixed drinking habits
* It is accompanied by intestinal diseases that seriously damage the intestinal barrier, such as inflammatory bowel disease, Crohn's disease, intestinal tuberculosis, ischemic bowel disease, radiation enteritis, and intestinal infectious diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale（PANSS）score | At the beginning of treatment, at 4 weeks and at the end of 8 weeks
  PANSS is a scale used to assess the psychotic symptoms of the client.This scale is evaluated by trained doctors, usually through conversation and observation, and scored after the examination. Score before and after treatment and during treatment can evaluate the severity of the disease and treatment effect.
Positive and Negative Syndrome Scale（PANSS）score | at the end of 4 weeks
  PANSS is a scale used to assess the psychotic symptoms of the client.This scale is evaluated by trained doctors, usually through conversation and observation, and scored after the examination. Score before and after treatment and during treatment can evaluate the severity of the disease and treatment effect.
Positive and Negative Syndrome Scale（PANSS）score | at the end of 8 weeks
  PANSS is a scale used to assess the psychotic symptoms of the client.This scale is evaluated by trained doctors, usually through conversation and observation, and scored after the examination. Score before and after treatment and during treatment can evaluate the severity of the disease and treatment effect.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Zhu, professor, Study Director — First Affiliated Hospital Xi'an Jiaotong University